CLINICAL TRIAL: NCT06081933
Title: Intranasal Dexmedetomidine Versus Intravenous Dexmedetomidine for Improving Quality of the Operative Field in Functional Endoscopic Sinus Surgery: A Randomized Triple-Blind Trial
Brief Title: Intranasal Dexmedetomidine Versus Intravenous Dexmedetomidine for Improving Quality of Endoscopic Sinus Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed Fouad Algyar, Lecturer of Anaesthesiology, Surgical Intensive Care and Pain Medicine, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MKSU-50-9-20
Record Dates: First submitted 2022-12-11; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-03

CONDITIONS: Dexmedetomidine; Functional Endoscopic Sinus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intranasal dexmedetomidine (Experimental): Patients will receive 1.5 micro g/kg intranasal dexmedetomidine diluted with saline + infusion saline
  Interventions: Drug: intranasal dexmedetomidine
- intravenous dexmedetomidine (Experimental): patients will receive 0.1- 0.4 micro g/kg intravenous infusion dexmedetomidine + intranasal saline.
  Interventions: Drug: intravenous dexmedetomidine

INTERVENTIONS:
Drug: intranasal dexmedetomidine — Patients will receive 1.5 micro g/kg intranasal dexmedetomidine diluted with saline + infusion saline
  Arms: intranasal dexmedetomidine
Drug: intravenous dexmedetomidine — patients will receive 0.1- 0.4 micro g/kg intravenous infusion dexmedetomidine + intranasal saline.
  Arms: intravenous dexmedetomidine

SUMMARY:
compare intranasal dexmedetomidine versus intravenous dexmedetomidine for improving quality of the operative field in Functional endoscopic sinus surgery

DETAILED DESCRIPTION:
Functional endoscopic sinus surgery is a well-established therapeutic option for intractable CRS and other indications. Functional endoscopic sinus surgery is a minimally invasive procedure and is commonly performed under controlled hypotensive anesthesia. In case of major bleeding, risk of complications such as meningitis, blindness, intracranial injury, cerebrospinal fluid leakage and the duration of surgery increase. Intraoperative bleeding is the most common factor that diminishes visibility, resulting in an increased incidence of complications.

Dexmedetomidine is a highly selective α2 adreno-receptor agonist with higher affinity to a2 adreno-receptor than clonidine, and this makes dexmedetomidine primarily sedative and anxiolytic.The elimination half-life of dexmedetomidine (t1/2b) is 2 h and the redistribution half-life (t1/2a) is 6 min, and this short half-life makes it an ideal drug for intravenous titration.

Intranasal Dexmedetomidine is convenient, effective, and noninvasive and also has useful analgesic and sedative effects in surgical procedures. Cheung's research has shown that intranasal Dexmedetomidine 1 and 1.5 micro/kg in surgical procedures produced significant sedation and less postoperative pain. Several previous research were determined the effect of intranasal dexmedetomidine in several clinical evaluations

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent Functional Endoscopic Sinus Surgery
* American Society of Anesthesiologists (ASA) physical status classification I or II

Exclusion Criteria:

* Patients with a body mass index > 30 kg/m2 existing or recent significant disease
* contraindications to the use of dexmedetomidine
* history or presence of a significant disease significant cardiovascular disease risk factors
* significant coronary artery disease or any known genetic predisposition
* history of any kind of drug allergy
* drug abuse
* psychological or other emotional problems
* special diet or lifestyle
* clinically significant abnormal findings in physical examination, electrocardiographic (ECG) or laboratory screening
* known systemic disease requiring the use of anticoagulants, patients with a history of previous Functional Endoscopic Sinus Surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Improving quality of the operative field | 24 hours postoperative
  Patients' satisfaction will be measured immediately postoperative and after 24 hours using a five-point Likert scale consisting of "very dissatisfied," "dissatisfied," "unsure," "satisfied," and "very satisfied.

SECONDARY OUTCOMES:
Heart rate will be evaluated | every 5 min till the end of procedure
  Heart rate will be recorded at baseline and every 5 min till the end of procedure
Mean arterial blood pressure will be evaluated. | every 5 min till the end of procedure
  Mean arterial blood pressure will be recorded at baseline and every 5 min till the end of procedure
Pain score will be evaluated. | 24 hour postoperatively
  Pain score will be evaluated measured with Numerical rating scale The numerical scale is most commonly 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable
Adverse reactions of hemostatic stuffing after FESS will be evaluated. | 24 hour postoperatively
  1=no swelling, can tolerate; 2= swelling, can barely tolerate; 3= swelling, cannot tolerate

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Ebeid, MD, Principal Investigator — Lecturer of Otorhinolaryngology, Faculty of medicine, Tanta University, Egypt
Locations (1):
- Mohammad Fouad Algyar, Kafr ash Shaykh, Kafr El-Shaikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the principal investigator
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After one year